CLINICAL TRIAL: NCT01806740
Title: Phase IV Study of DCE-MRI Using Dotarem® in Evaluation of Therapeutic Response to Sorafenib in Patients With Advanced Stage HCC
Brief Title: DCE-MRI Using Dotarem® in Evaluation of Therapeutic Response to Sorafenib in Patients With Advanced Stage HCC
Acronym: DCE-MRI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The planned number of enrolled patients was not reached.
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-057
Record Dates: First submitted 2012-11-06; First posted 2013-03-07 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: DCE-MRI; Sorafenib response
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadoterate meglumine (Experimental): there is one single arm of patients (no comparative arm)
  Interventions: Drug: Gadoterate meglumine

INTERVENTIONS:
Drug: Gadoterate meglumine — Gadoterate meglumine was administered at a dose of 0.1 mmol/kg (0.2 mL/kg) using a power injector, in an intravenous bolus at a rate of 3 mL/sec.
  Other Names: gadoteric acid; Dotarem

SUMMARY:
The main objective is to evaluate the value of dynamic contrast-enhanced Magnetic Resonance Imaging (DCE-MRI) in prediction of response of patients with hepatocellular carcinoma (HCC) to treatment with Sorafenib assessed by mRECIST.

DETAILED DESCRIPTION:
One of the secondary objectives was to evaluate the correlation between DCE-MRI perfusion parameters at baseline and:

* Overall Survival (OS)
* Progression-Free Survival (PFS)
* Time to Progression (TTP)

Three DCE-MRI examinations were done during the study:

* at the enrolment and initiation of the sorafenib treatment
* one week after initiation of the sorafenib treatment
* two weeks after initiation of the sorafenib treatment

DCE-MRI perfusion parameters were assessed by a centralized radiologist at baseline (corresponding to the day of enrolment and initiation of Sorafenib treatment), week 1 and week 2.

According to mRECIST criteria, HCC lesions were evaluated on computed tomography images by two on-site radiologists at the time of enrolment and 8 weeks later (2 months). OS, PFS and TTP were calculated from survival and tumor progression data recorded one year after initiation of the sorafenib treatment.

ELIGIBILITY:
1. Male and female adult patients (age ≥ 20 years old)
2. Patients diagnosed with unresectable HCC [Child Pugh class A and major vascular invasion, extrahapatic metastasis, or progression after transarterial chemoembolization more than 2 times]
3. Presence of mRECIST target lesion within liver [lesion which can be classified as a RECIST measurable lesion (can be measured ≥ 1 cm in at least one dimension), lesion suitable for repeated measure, lesion showing intraluminal arterial enhancement on contrast-enhanced CT or MRI]
4. Patients planned to be treated with sorafenib
5. Patient with liver CT performed or planned to be performed within 4 weeks before initiation of sorafenib treatment
6. Patient with a life expectancy of 12 weeks or more
7. No previous treatment with sorafenib
8. Female patients who are surgically sterilized, or post-menopausal (minimum 12 months of amenorrhea) or who have a documented negative urine hCG test at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05-09 (Actual); Primary Completion 2015-10-12 (Actual); Study Completion 2015-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Guerbet Korea, Seoul, Gangnam Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided after study completion.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Despite several extensions of the recruitment period, the planned number of enrolled patients was still not reached after 2 years and the study was prematurely discontinued.
  A total of 37 patients were enrolled in four study sites.
Groups:
- Gadoterate Meglumine: All patients who received gadoterate meglumine.
Period: Overall Study
Arm/Group | Gadoterate Meglumine
Started | 37
Completed | 31
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Patient's refusal of treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gadoterate Meglumine
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.06 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 60.03 (9.17)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between DCE-MRI Perfusion Parameters and the Response of Target Lesions to Sorafenib
Description: To evaluate the correlation between DCE-MRI perfusion parameters (Ktrans, AUC, ve, kep, T1, Wash-in, Washout) at baseline, week 1 and week 2, and the response of target lesions to sorafenib.
  * Ktrans: volume transfer constant between blood plasma and extravascular extracellular space
  * AUC : area under the curve of tissue gadolinium concentration-time
  * ve: fractional volume of extravascular extracellular space
  * kep: rate constant between extravascular extracellular space and blood plasma (=Ktrans/ve)
  * T1: longitudinal relaxation time
  * Wash-in: slope of the early enhancement curve
  * Washout: slope of the late enhancement curve
  The response of target lesions was assessed by mRECIST at 2 months after initiation of treatment (sorafenib).
  The correlation analyses were done using Pearson or Spearman correlation coefficient.
Time Frame: 3 months
Population: A total of 26 target lesions were identified in the 15 patients of the full analysis set (patients with available data for the primary criteria). One lesion was not assessed at baseline, week 1 and week 2 for all parameters and one lesion was not assessed at baseline and week 1 for Ktrans, ve and kep.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Target lesions
Groups:
- Baseline: DCE-MRI perfusion parameters assessed at baseline (initiation of the sorafenib treatment)
- Week 1: DCE-MRI perfusion parameters assessed one week after initiation of the sorafenib treatment
- Week 2: DCE-MRI perfusion parameters assessed two weeks after initiation of the sorafenib treatment
Arm/Group | Baseline | Week 1 | Week 2
Number analyzed (Participants) | 15 | 15 | 15
Number analyzed (Target lesions) | 25 | 25 | 25
correlation coefficient
  Ktrans (mean): number analyzed (Target lesions) | 24 | 24 | 25
  Ktrans (mean) | -0.29 | -0.38 | -0.38
  AUC (mean) | -0.53 | -0.60 | -0.62
  ve (mean): number analyzed (Target lesions) | 24 | 24 | 25
  ve (mean) | -0.19 | -0.33 | -0.34
  kep (mean): number analyzed (Target lesions) | 24 | 24 | 25
  kep (mean) | -0.07 | -0.24 | -0.17
  T1 (mean) | 0.05 | 0.30 | 0.18
  Wash-in (mean) | -0.42 | -0.48 | -0.52
  Washout (mean) | -0.31 | -0.48 | -0.36

2. Secondary Outcome: Correlation Coefficient Between DCE-MRI Perfusion Parameters at Baseline and Overall Survival
Description: To evaluate the correlation between DCE-MRI perfusion parameters (Ktrans, AUC, ve, kep, T1, wash-in, washout) at baseline and overall survival.
  The overall survival was calculated from the patient's survival status recorded one year after initiation of the sorafenib treatment.
  The correlation analyses were done using Pearson or Spearman correlation coefficient.
Time Frame: 1 year
Population: Among the 15 patients of the full analysis set (26 target lesions), one patient was lost to follow-up. Consequently, 14 patients had data for overall survival (23 target lesions). One lesion was not assessed for Ktrans, ve and kep.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Target lesions
Groups:
- Baseline: DCE-MRI perfusion parameters assessed at baseline (initiation of sorafenib treatment)
Arm/Group | Baseline
Number analyzed (Participants) | 14
Number analyzed (Target lesions) | 23
correlation coefficient
  Ktrans (mean): number analyzed (Target lesions) | 22
  Ktrans (mean) | 0.09
  AUC (mean) | -0.08
  ve (mean): number analyzed (Target lesions) | 22
  ve (mean) | 0.35
  kep (mean): number analyzed (Target lesions) | 22
  kep (mean) | -0.05
  T1 (mean) | -0.14
  Wash-in (mean) | -0.02
  Washout (mean) | -0.04

3. Secondary Outcome: Correlation Coefficient Between DCE-MRI Perfusion Parameters at Baseline and Progression Free Survival
Description: To evaluate the correlation between DCE-MRI perfusion parameters (Ktrans, AUC, ve, kep, T1, wash-in, washout) at baseline and progression free survival.
  The progression free survival was calculated from the patient's survival status and tumor progression status recorded one year after initiation of the sorafenib treatment.
  The correlation analyses were done using Pearson or Spearman correlation coefficient.
Time Frame: 1 year
Population: Among the 15 patients of the full analysis set (26 target lesions), 13 had data for progression free survival (22 target lesions). One lesion was not assessed for Ktrans, ve and kep.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Target lesions
Arm/Group | Baseline
Number analyzed (Participants) | 13
Number analyzed (Target lesions) | 22
correlation coefficient
  Ktrans (mean): number analyzed (Target lesions) | 21
  Ktrans (mean) | -0.24
  AUC (mean) | -0.45
  ve (mean): number analyzed (Target lesions) | 21
  ve (mean) | 0.17
  kep (mean): number analyzed (Target lesions) | 21
  kep (mean) | -0.23
  T1 (mean) | -0.15
  Wash-in (mean) | -0.31
  Washout (mean) | -0.29

4. Secondary Outcome: Correlation Coefficient Between DCE-MRI Perfusion Parameters at Baseline and Time to Progression
Description: To evaluate the correlation between DCE-MRI perfusion parameters (Ktrans, AUC, ve, kep, T1, wash-in, washout) at baseline and time to progression.
  The time to progression was calculated from the patient's survival status and tumor progression status recorded one year after initiation of the sorafenib treatment.
  The correlation analyses were done using Pearson or Spearman correlation coefficient.
Time Frame: 1 year
Population: Among the 15 patients of the full analysis set (26 target lesions), 4 patients had data for time to progression (7 target lesions).
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Target lesions
Arm/Group | Baseline
Number analyzed (Participants) | 4
Number analyzed (Target lesions) | 7
correlation coefficient
  Ktrans (mean) | -0.72
  AUC (mean) | -0.64
  ve (mean) | -0.68
  kep (mean) | -0.17
  T1 (mean) | 0.24
  Wash-in (mean) | -0.70
  Washout (mean) | -0.42

ADVERSE EVENTS:
Time Frame: 3 months (from the informed consent signature to 2 months after initiation of the sorafenib treatment)
Arm/Group | Gadoterate Meglumine
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 7/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadoterate Meglumine (N=31)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadoterate Meglumine (N=31)
Diarrhoea (Gastrointestinal disorders) | 10 (11)
Nausea (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Blood pressure increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Penile erythema (Reproductive system and breast disorders) | 1 (1)
Penile oedema (Reproductive system and breast disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The small number of patients included and analyzed was a major limitation to interpret the efficacy results, inducing high variability in DCE-MRI perfusion parameters, OS, PFS and TTP values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other